CLINICAL TRIAL: NCT05563558
Title: A Phase 2 Clinical Trial of Pembrolizumab in Combination With Carboplatin and Cabazitaxel in Aggressive Variant Metastatic Castration Resistant Prostate Cancer
Brief Title: Pembrolizumab, Carboplatin and Cabazitaxel in Aggressive Metastatic Castration Resistant Prostate Cancer (PEAPOD_FOS)
Acronym: PEAPOD_FOS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Oncosur (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEAPOD_FOS04/2022
Record Dates: First submitted 2022-09-21; First posted 2022-10-03 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — pembrolizumab; Carboplatin; cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): 6 cycles of Pembrolizumab+Cabazitaxel+Carboplatin + 15 cycles of Pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cabazitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Included in arm/group description
Drug: Carboplatin — Included in arm/group description
Drug: Cabazitaxel — Included in arm/group description

SUMMARY:
It is a Phase 2 clinical trial of Pembrolizumab in combination with Carboplatin and Cabazitaxel in Aggressive Variant Metastatic Castration Resistant Prostate Cancer.

It is divided into two parts: an induction period of 6 cycles of 3 weeks each cycle of Pembrolizumab+Cabazitaxel+Carboplatino and a maintenance phase of 15 cycles of 6 weeks each cycle of Pembrolizumab.

DETAILED DESCRIPTION:
Aggressive variant prostate cancer is a clinically defined subset of metastatic castration resistant prostate cancers characterized by the absence of response to AR targeted agents and neuroendocrine features. The treatments that are currently available are not effective and represent an unmet clinical need. This subgroup has been molecularly characterized and associate loss of key tumor suppressors, including TP53, PTEN and RB, and neuroendocrine features. Carboplatin and cabazitaxel have demonstrated promising activity in this scenario although virtually all patients succumb to the disease. Pembrolizumab has demonstrated activity in neuroendocrine tumors. In this trial will be evaluated the activity and safety of pembrolizumab in combination with the most active chemotherapy regiment available to date in aggressive variant prostate cancer, carboplatin plus cabazitaxel

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are at least 18 years of age on the day of signing informed consent
* Histologically confirmed diagnosis of adenocarcinoma and/or neuroendocrine carcinoma of the prostate will be enrolled in this study
* Presence of metastatic disease documented on imaging studies (bone scan, computed tomography (CT) and/or magnetic resonance imaging (MRI) scans
* At least one of the following Aggressive Variant Prostate Cancer (AVPC) Criteria

  1. Histologically proven small cell (neuroendocrine) prostate cancer
  2. Exclusive visceral metastases
  3. Predominantly lytic bone metastases
  4. Bulky lymph nodes (≥ 5 cm in longest dimension) or high-grade pelvic/prostatic masses
  5. Low PSA (≤10 ng/ml) at initial presentation in the presence of extensive disease (≥20 metastases)
  6. Elevated serum Lactate Dehydrogenase (LDH) (≥2 x ULN) or carcinoembryonic antigen (CEA) (≥2 x Upper limit (UL))
  7. Short time to castration-resistance (≤6 months).
* Male participants: a male participant must agree to use a contraception as detailed in Appendix 3 of the protocol during the treatment period and for at least after the last dose of study treatment and refrain from donating sperm during this period
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have provided archival tumor tissue sample obtained in the previous year since or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
* Have adequate organ function as defined in the table 1 of the protocol. Specimens must be collected within 10 days prior to the start of study intervention.
* Criteria for known Hepatitis B (HBV) and C (HCV) positive subjects

  1. Hepatitis B and C screening tests are not required unless:

     * Known history of HBV or HCV infection
     * As mandated by local health authority
  2. Hepatitis B positive subjects

     * Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
     * Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
  3. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening. • Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., Cytotoxic T-Lymphocyte Antigen 4 (CTLA-4), OX-40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to informed consent signature.
* Has received previous treatment with cabazitaxel or carboplatin.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (non-CNS) disease.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, carboplatin or cabazitaxel and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy
* Has congestive Heart failure New York Heart Association (NYHA) ≥2.
* Has hypoacusis grade ≥2.
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

Note: Hepatitis B and C screening tests are not required unless:

* Known history of HBV and HCV infection
* As mandated by local health authority

  * Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
  * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  * Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events | through study completion, an average of 2 years
  Incidence of adverse events (AEs) graded according to NCI-CTCAE v 5.0 criteria
Efficacy - Radiographic Progression-Free Survival rate | 6 months
  To assess the safety of pembrolizumab in combination with carboplatin and cabazitaxel according to 6 months Radiographic Progression-Free Survival rate (rPFS) according to the Prostate Cancer Working Group 3 (PCWG3 ).

SECONDARY OUTCOMES:
Efficacy - Progression Free-Survival | 12 months
  To determine radiographic Progression Free-Survival at 12 months
Efficacy - Response rate | through study completion, an average of 2 years
  To evaluate response rate by Prostate Cancer Working Group (PCWG) modified RECIST 1.1
Efficacy - PSA response | through study completion, an average of 2 years
  To evaluate PSA response (when PSA is evaluable)
Efficacy - PSA progression-free survival | through study completion, an average of 2 years
  To determine PSA progression-free survival (PSA-PFS)
Efficacy - progression-free survival | through study completion, an average of 2 years
  To determine progression-free survival (PFS)
Efficacy - overall survival | through study completion, an average of 2 years
  To determine overall survival (OS)

OTHER OUTCOMES:
Exploratory objective - Correlation of efficacy endpoints with AVPC- Molecular-Classification (MC) | through study completion, an average of 2 years
  Correlation of efficacy endpoints with AVPC- Molecular-Classification (MC) defined as the presence of tumour mutations in two of the following genes: P53, phosphatase and tensin homolog (PTEN) or Retinoblastoma (RB).
Exploratory objective - Correlation of efficacy endpoints with neuroendocrine signature | through study completion, an average of 2 years
  Correlation of efficacy endpoints with neuroendocrine signature in the Circulating tumor DNA (ctDNA) methylation pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Gonzalez-Billalabeitia, Dr, Principal Investigator — Hospital Universitario 12 de Octubre, Madrid; Teresa Alonso Gordoa, Dr, Principal Investigator — Hospital Universitario Ramón y Cajal; Álvaro Pinto Marín, Dr, Principal Investigator — Hospital Universitario La Paz; Ignacio Durán Martínez, Dr, Principal Investigator — Hospital Universitario Marqués de Valdecilla; Begoña Mellado González, Dr, Principal Investigator — Hospital Clinic of Barcelona; David Lorente Estellés, Dr, Principal Investigator — Hospital Provincial De Castellón; Albert Font Pous, Dr, Principal Investigator — ICO- Badalona; Sergio Vazquez Estévez, Dr, Principal Investigator — Hospital Lucus Augusti; Javier Puente, Dr, Principal Investigator — Hospital San Carlos, Madrid
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain